CLINICAL TRIAL: NCT00929370
Title: A 4-Part Parallel Group, Randomized, Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Repeat Doses of GSK1018921 in Healthy Volunteers and Stable Patients With Schizophrenia and to Evaluate Its Effects on Pharmacokinetics of Midazolam.
Brief Title: A Repeat Dose Study With GSK1018921 to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics in Healthy Volunteers and Patients With Schizophrenia and to Evaluate Its Effect on PK of Midazolam.
Acronym: GT1110791
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has now been terminated due to changes in project strategy. Current available data will be analysed and reported in a synoptic study report.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110791
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; GSK1018921; GlyT-1 inhibitor; Healthy Volunteers; CSF; Patient; Midazolam
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- GSK1018921 (Experimental): Glycine Transporter-1 inhibitor to modulate the NMDA receptor.
  Interventions: Drug: Glycine Transporter-1 inhibitor

INTERVENTIONS:
Drug: Glycine Transporter-1 inhibitor — GSK1018921 is a potent and selective inhibitor of the glycine transporter-1 (GlyT-1).

SUMMARY:
The purpose of this study is to understand safety and tolerability of the drug GSK1018921 after 14 days of dosing in healthy volunteers and then in patient volunteers.

DETAILED DESCRIPTION:
This is a four part, parallel group, randomised, study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) effects of repeat doses of GSK1018921 in healthy volunteers and stable patients with schizophrenia and to evaluate its effect on pharmacokinetics of midazolam. Part A will evaluate 14 days repeat BID dosing in at least three cohorts of healthy volunteers, to assess safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK1018921. Part B will study the potential drug interaction of GSK1018921 (Maximum Tolerated Dose from Part A) with midazolam with 14 days repeat BID dosing in healthy volunteers and therefore will assess the PK, safety and tolerability. Part C will be a single dose study in healthy volunteers and will include CSF sampling to assess the concentration of GSK1018921 and glycine in CSF with two doses (80 and 200 mg). Part D will study stable patients with schizophrenia, to assess safety, tolerability, PK and PD following 28 days of repeat BID dosing.

Safety assessments will include physical examination, 12-lead ECGs, holter monitoring, vital signs, orthostatic vital signs, visual assessments, and clinical lab test. Tolerability will be assessed by collecting Adverse Events.

PD assessments will include glycine in red blood cells, plasma and CSF, as well as CogState Battery test, Visual Assessment Scale, Positive And Negative Symptom Scores (PANSS) and Clinical Global Impression scales of change.

ELIGIBILITY:
All subjects (Healthy and Patients)

Exclusion Criteria:

* History of drug or alcohol abuse.
* Consumption of drug, food or drink affecting the CYP450 metabolism pathway.
* Has received investigational drug within 30 days to 5 half lives or twice the duration of the biological effect of any drug (which ever is the longer).
* Donation of blood in excess of 500mL within a 56 day period.

Patients eligibility

- Stable patients with schizophrenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and tolerability endpoints consisting of: adverse events; 12-lead ECG; vital signs, clinical laboratory evaluations and PK parameters. | 14 days twice daily dosing.
Part B: Midazolam PK following single and repeat doses of GSK1018921. | 14 days twice daily dosing.
Part C: Plasma & CSF glycine concentrations following single doses og GSK1018921. | After single dosing.
Part D: Safety and tolerability endpoints consisting of: adverse events; 12-lead ECG; vital signs, clinical laboratory evaluations and movement scales Simpson Angus Scale, AIMS and Barnes akathisia Scale. | 28 days

SECONDARY OUTCOMES:
Part A: Effects of GSK1018921 on VAS | 14 days.
Part B: None | 0
Part C: GSK1018921 plasma exposure-CSF glycine relationship | After single dosing.
Part D: Effects of GSK1018921 on VAS, PANSS and CGI | 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Bellaire, Texas